CLINICAL TRIAL: NCT00604773
Title: Incidence of Delirium in Critically Ill Patients in a Dutch University Hospital
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: M. van den Boogaard, MSc, RN, CCRN, Radboud University Nijmegen Medical Centre
Other Study IDs: Radboud 2007/283
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2009-02

CONDITIONS: Delirium
Keywords: delirium; critical care; risk factors; prediction
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- delirious patients: minimal one positive CAM-ICU score during ICU admission
- non-delirious patients: without any positive CAM-ICU scores during ICU admission

SUMMARY:
The objective of this study is to determine the incidence of delirium in adults patients who are admitted at the critical care unit of a Dutch University Hospital.

The primary aim is to determine the incidence of delirium and to determine risk factors for this group of patients to develop a prediction model.

A secondary aim is to find differences between delirious patients and non-delirious patients on different aspects of diagnostics, treatment and care, outcome, length of stay, and inflammation.

According to Dutch law, the need to obtain informed consent was waived by the Committee on Research Involving Human Subjects (CMO) of Nijmegen for this observational study (2007/283).

ELIGIBILITY:
Inclusion Criteria:

* all adult patients (18 years and older) admitted at the critical care unit of our hospital

Exclusion Criteria:

* not able to understand Dutch
* patients with serious hearing and visibility disabilities
* mentally retarded patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
delirium | during admission at the critical care

SECONDARY OUTCOMES:
markers of inflammation | within 24 hours of delirium diagnosis
biomarkers | within 24 hours of delirium diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Hans vd Hoeven, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Critical Care, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] van den Boogaard M, Pickkers P, Slooter AJ, Kuiper MA, Spronk PE, van der Voort PH, van der Hoeven JG, Donders R, van Achterberg T, Schoonhoven L. Development and validation of PRE-DELIRIC (PREdiction of DELIRium in ICu patients) delirium prediction model for intensive care patients: observational multicentre study. BMJ. 2012 Feb 9;344:e420. doi: 10.1136/bmj.e420. PMID 22323509
- [Derived] van den Boogaard M, Kox M, Quinn KL, van Achterberg T, van der Hoeven JG, Schoonhoven L, Pickkers P. Biomarkers associated with delirium in critically ill patients and their relation with long-term subjective cognitive dysfunction; indications for different pathways governing delirium in inflamed and noninflamed patients. Crit Care. 2011;15(6):R297. doi: 10.1186/cc10598. Epub 2011 Dec 29. PMID 22206727
- [Derived] van den Boogaard M, van Swelm RP, Russel FG, Heemskerk S, van der Hoeven JG, Masereeuw R, Pickkers P. Urinary protein profiling in hyperactive delirium and non-delirium cardiac surgery ICU patients. Proteome Sci. 2011 Mar 22;9:13. doi: 10.1186/1477-5956-9-13. PMID 21426560